CLINICAL TRIAL: NCT01160185
Title: Meta-analysis of Efficacy of Topotecan and Other Treatments for Recurrent Carcinoma of the Cervix
Brief Title: Meta-analysis of Efficacy of Topotecan
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Study Director, GSK
Other Study IDs: 114015
Record Dates: First submitted 2010-07-08; First posted 2010-07-12 (Estimated); Last update posted 2010-07-12 (Estimated); Status verified 2010-07

CONDITIONS: Cervical Intraepithelial Neoplasia
MeSH Terms: conditions — Uterine Cervical Dysplasia | interventions — Paclitaxel; Cisplatin; Topotecan

STUDY DESIGN:
Time Perspective: Retrospective

GROUPS / COHORTS (3):
- cisplatin
  Interventions: Drug: cisplatin
- cisplatin + topotecan
  Interventions: Drug: cisplatin; Drug: topotecan
- cisplatin + paclitaxel
  Interventions: Drug: paclitaxel; Drug: cisplatin

INTERVENTIONS:
Drug: paclitaxel — paclitacel
  Groups: cisplatin + paclitaxel
Drug: cisplatin — cisplatin monotherapy
Drug: topotecan — topotecan
  Groups: cisplatin + topotecan

SUMMARY:
This meta-analysis was conducted to investigate the efficacy of Topotecan and other treatments for recurrent and stage IVB carcinoma of the cervix

DETAILED DESCRIPTION:
Studies included in the meta-analysis were: GOG-0179, GOG-0204 & GOG-0169

ELIGIBILITY:
Inclusion Criteria:

* Randomised Clinical Trials or systematic reviews or meta-analyses
* Treatment with topotecan or platinum-based single and combination regimens in female patients of any race with cancer of the cervix recurrent after radiotherapy or stage IVB disease

Exclusion Criteria:

* None

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The search was designed to identify all clinical data published since the Cancer Care Ontario systematic review in 2006. The Cancer Care Ontario systematic review searched MEDLINE (1966 to February 2006), EMBASE (1980 to February 2006), the Cochrane Library (Cochrane Database of Systematic Reviews (2006 Issue 1), and Cochrane Controlled Trials Register (2006 Issue 1)), the Canadian Medical Association Infobase, and the National Guidelines Clearinghouse. The conference proceedings of the American Society of Clinical Oncology (1995-2005) and the European Society of Medical Oncology (2002-2005) were also searched. The search was conducted on 18 December 2008.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2009-06; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Survival | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline